CLINICAL TRIAL: NCT05862142
Title: A Predictive Model for Oropharyngeal Dysphagia in Non-hospitalized Older Patients: Building Bridges Between Detection and Decision-making
Brief Title: A Predictive Model for Oropharyngeal Dysphagia in Non-hospitalized Older Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-DOF-2022-121
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Deglutition Disorders; Otorhinolaryngologic Diseases; Oropharyngeal Dysphagia
Keywords: Older people; Predictive models
MeSH Terms: conditions — Deglutition Disorders; Otorhinolaryngologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Oropharyngeal dysphagia (OD) is a highly prevalent and growing condition in the older population. It affects approximately one in three community-dwelling elderly, almost half of the geriatric patients, and even more than half of elderly nursing home residents.

The main complications of OD are respiratory infections such as aspiration pneumonia, malnutrition, and dehydration. It supposes substantial costs for the healthcare system, increases the risk for (re)admissions and length of stay, and has an important impact on the quality of life of people who suffer from it.

The aim of this study is to develop a predictive model to identify non-hospitalized older patients at risk for oropharyngeal dysphagia, quantify that risk, and facilitate decision-making according to personal, clinical, and socio-emotional characteristics.

DETAILED DESCRIPTION:
Given the high prevalence of Oropharyngeal Dysphagia (OD) in older people and the difficulty to detect it, the investigators purpose to develop a predictive model to identify non-hospitalized older patients at risk for OD, quantify that risk, and facilitate decision-making.

Objectives:

Main objective:

- Develop a predictive model for oropharyngeal dysphagia in non-hospitalized older patients (≥ 65 years).

Secondary objectives:

* Identify predictive factors for OD among the studied population.
* Contribute to the characterization of OD in older people through a retrospective analysis of videofluoroscopic studies and clinical evaluations.
* Define different models of intervention from a multidimensional approach.

ELIGIBILITY:
Inclusion Criteria:

* Older people between 65 and 99 years.
* Swallowing assessed with Videofluoroscopy
* Non-hospitalized patients (swallowing assessed on an outpatient basis)

Exclusion Criteria:

* There are no exclusion criteria in relation to the gender or ethnicity of the participants. Failure to meet one of the inclusion criteria will result in the participant's exclusion from the study sample.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older patients (≥ 65 years) referred to the Physical Medicine and Rehabilitation Service of Hospital de la Santa Creu i Sant Pau for a swallowing study between 2015 and 2023.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-06 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Dysphagia Outcome and Severity Scale (DOSS). Instrumental assessment tool used: Videofluoroscopic Swallowing study (VFSS) | Up to 8 years
  It is a simple, easy-to-use, 7-point scale developed to systematically rate the functional severity of dysphagia based on objective assessment and make recommendations for diet level, independence level, and type of nutrition Range: 1 Nothing by mouth (NPO) - 7 Full oral intake, normal.
Penetration Aspiration Scale (PAS). Instrumental assessment tool used: Videofluoroscopic Swallowing study (VFSS) | Up to 8 years
  It is a is a rank ordered scale that classifies the depth of penetrated or aspirated material and the patient's response to airway invasion. Range: 1 No airway penetration - 8 Airway aspiration, no cough.
Bolus Residue Scale (BRS). Instrumental assessment tool used: Videofluoroscopic Swallowing study (VFSS) | Up to 8 years
  It is a simple, easy-to-carry-out, and accessible analysis method to rate and locate pharyngeal retention. Range: 1 No residue - 6 Residue in valleculae and posterior pharyngeal wall and piriform sinus.
Functional Oral Intake Scale (FOIS). Instrumental assessment tool used: Videofluoroscopic Swallowing study (VFSS) | Up to 8 years
  It is a reliable and valid tool to assess functional oral intake of food and liquids in patients with oropharyngeal dysphagia (OD). Range: 1 Nothing by mouth (NPO) - 7 Full oral intake without restrictions.

SECONDARY OUTCOMES:
Predictive value of pharyngeal width at rest for aspiration (JOSCYL width). Instrumental assessment tool used: Videofluoroscopic Swallowing study (VFSS) | Up to 8 years
  The JOSCYL Width Scale is calculated by averaging two pharyngeal widths: 1) lower margin of the mandible to C2 and 2) epiglottis to C3.